CLINICAL TRIAL: NCT02114671
Title: A Randomised, Assessor-blind, Placebo and Active Controlled, Parallel Group Study to Assess the Phototoxic Potential of Faldaprevir (Administered Orally, Once Daily) for 6 Days in Healthy Male and Female Subjects
Brief Title: A Study to Investigate the Phototoxic Potential of Faldaprevir
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1241.42; 2013-000767-88 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — faldaprevir; Ciprofloxacin

ARMS (4):
- Faldaprevir QD high dose (Experimental): capsules, oral administration with 240 ml water, fed conditions
  Interventions: Drug: Faldaprevir high dose
- Faldaprevir QD low dose (Experimental): tablets/capsules, oral administration with 240 ml water, fed conditions
  Interventions: Drug: Faldaprevir low dose
- Placebo (Placebo Comparator): capsules, oral administration with 240 ml water, fed conditions
  Interventions: Drug: Placebo
- Ciprofloxacin (Active Comparator): tablets, oral administration with 240 ml water, fed conditions
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Faldaprevir high dose — capsules, oral
  Arms: Faldaprevir QD high dose
Drug: Placebo — capsule, oral
  Arms: Placebo
Drug: Ciprofloxacin — tablets, oral
  Arms: Ciprofloxacin
Drug: Faldaprevir low dose — capsules, oral
  Arms: Faldaprevir QD low dose

SUMMARY:
To investigate the potential of Faldaprevir to induce skin phototoxicity, immediate or delayed type, to UV light and visible light in healthy male and female subjects. To investigate the degree, wavelength dependency, severity, pigmentation and morphology of the phototoxic effects. The persistence of the phototoxic susceptibility will be explored following cessation of study medication. Within a sunscreen sub-study, the efficacy of commercially available high factor sunscreen will also be assessed in terms of its potential to prevent any phototoxic skin responses seen. The safety and tolerability of Faldaprevir will also be assessed.

ELIGIBILITY:
Inclusion criteria:

* Health male and female subjects with no clinically significant abnormality (according to the Investigator's assessment) identified from a complete medical history, physical examination, whole body skin assessment, 12-lead ECG, vital signs and clinical laboratory tests. In particular, there should be no evidence of abnormal photosensitivity
* Sun-reactive skin phototype I, II, or III

Exclusion criteria:

- Any relevant deviation from healthy conditions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with drug related adverse events | 17 days
Change in minimum erythema dose (MED) at each wavelength tested, before and during treatment. The change will be quantified by the phototoxic index at 24 hrs (delayed erythema) derived by dividing the baseline MED by that during treatment | 7 days
Percentage of subjects with drug related adverse events | 17 days

SECONDARY OUTCOMES:
Degree of phototoxic effects by phototoxic index | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.42.44001 Boehringer Ingelheim Investigational Site, Edinburgh, United Kingdom